CLINICAL TRIAL: NCT06288386
Title: Impact of Dental Composite Viscosity on Attachment Accuracy: a Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-ATTACHMENTS
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher filler content composite (Experimental): Attachments will be performed with a higher filler content flowable composite resin.
  Interventions: Device: GrandioSO Heavy Flow
- Lower filler content composite (Active Comparator): Attachments will be performed with a lower filler content flowable composite resin.
  Interventions: Device: Filtek Z350XT Flowable

INTERVENTIONS:
Device: GrandioSO Heavy Flow — Attachment will be performed with GrandioSO Heavy Flow.
  Arms: Higher filler content composite
Device: Filtek Z350XT Flowable — Attachment will be performed with Filtek Z350XT Flowable.
  Arms: Lower filler content composite

SUMMARY:
The present study will be a single-center, split-mouth, randomized controlled clinical trial. Patients undergoing orthodontic treatment with Invisalign aligners will be enrolled after signing the informed consent. Two different flowable composite resins will be evaluated for the performing of attachments using a split-mouth design:

* group A: Filtek Supreme Flow (3M Unitek, Monrovia, Calif)
* group B: Grandioso Heavy Flow (VOCO GmbH, Cuxhaven Germany)

Digital impressions with iTero intraoral scanner will be performed. The resulting 3D images will be superimposed onto the reference STL model, representing the pre- planned ideal attachment configuration. Digital scans will be used to assess any changes in shape of the attachments. Each tooth will be separated from the others and superimpositions of the single tooth will be performed with ZEISS Inspect software.

DETAILED DESCRIPTION:
The present study will be a single-center, split-mouth, randomized controlled clinical trial. Patients willing to start Invisalign treatment or refinement phases will be recruited from the Unit of Orthodontics and Pediatric Dentistry, Section of Dentistry, Department of Clinical, Surgical, Diagnostic and Pediatric Sciences, University of Pavia, Pavia, Italy. Each patient will sign the informed consent before participation. The bonding procedure will be the following: isolation of the working field with the placement of a cheek retractor, enamel etching with 37% orthophosphoric acid, rinsing and drying, application of a thin layer of ScotchBond adhesive (3M Unitek, Monrovia, Calif) and light curing. Then, patient will be divided into groups A and B: in group A, attachments will be realized using Filtek Supreme Flow (3M Unitek, Monrovia, Calif) for teeth belonging to mandibular left and maxillary right quadrants, whereas in the remaining quadrants, they will be realized using Grandioso Heavy Flow (VOCO GmbH, Cuxhaven Germany. In group B, quadrants will be inverted. After the bonding of the attachments, digital impressions with iTero intraoral scanner will be performed. The resulting 3D images will be superimposed onto the reference STL model, representing the pre-planned ideal attachment configuration. Digital scans will be used to assess any changes in shape of the attachments. Each tooth will be separated from the others and superimpositions of the single tooth will be performed with ZEISS Inspect software. For each of the five attachment surfaces the values obtained for the two composite resins will be compared using three key parameters: total mean discrepancy, mean of positive values only, and mean of negative values only. The analysis will be performed using R software, calculating descriptive statistics for each variable, including mean, standard deviation, median, minimum, and maximum values for each group. The normality of the distributions will be assessed using the Kolmogorov-Smirnov test. Subsequently, a t-test will be applied for inferential analysis of each variable.

For all tests, statistical significance will be set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing Invisalign orthodontic treatment

Exclusion Criteria:

* enamel demineralizations

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Changes in the shape of attachments | Baseline
  The shape changes of attachments will be evaluated through ZEISS Inspect software.
Change in excess of attachments | Baseline
  The excess of attachments will be evaluated through ZEISS Inspect software.
Change in defect of attachments | Baseline
  The defect of attachments will be evaluated through ZEISS Inspect software.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.